CLINICAL TRIAL: NCT01896609
Title: A Single Center, Prospective Phase IV, Open-Label, Randomized Trial Comparing the Efficacy , Tolerability, and Safety of Quadritherapy Regimen (Reiferon Retard® + Ribavirin + Nitazoxanide + Alfacalcidol ( Bon-One ®) ) Versus Triple Therapy Regimen (Reiferon Retard® + Ribavirin + Nitazoxanide) Versus the Standard of Care Regimen(Reiferon Retard® + Ribavirin) in the Treatment of Naïve Chronic Hepatitis- C Among the Egyptian Population. Effectiveness Will be Evaluated Based on Sustained Viral Response (SVR)
Brief Title: Trial Comparing the Efficacy, Tolerability and Safety Between Three Arms in Treatment of HCV in Egyptian Population
Acronym: Quadritherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MinaPharm Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV05012012
Record Dates: First submitted 2013-06-19; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Hepatitis c
Keywords: Chronic hepatitis c; Egyptian population; Reiferon Retard; Ribavirin; Nitazoxanide; Bon one
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; nitazoxanide; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Standard therpy) (Experimental): Arm 1 : subject randomized to this arm will be receiving the standard care therapy for 48 weeks:
  * Reiferon Retard® 160 µg /week subcutaneous injection.
  * Ribavirin in a dose of 13 mg/kg/day orally
  Interventions: Biological: Reiferon Retard in Arm 1; Drug: Ribavirin in Arm 1
- Arm 2 ( Xerovirinc) (Experimental): Arm 2 : Subjects randomized to this arm will be receiving the following medications for 48 weeks;
  * Reiferon Retard® 160 µg /week subcutaneous injection
  * Ribavirin in a dose of 13 mg/kg/day orally
  * Xerovirinc® 500mg twice daily orally.
  Interventions: Biological: Reiferon Retard in Arm 1; Drug: Xerovirinc in Arm 2; Drug: Ribavirin in Arm 1
- Arm 3 ( Bon one ) (Experimental): Arm 3: Subjects randomized to this arm will be receiving the following medications for 48 weeks:
  * Bon-One ® 0.5 µg daily orally
  * Reiferon Retard® 160 µg /week subcutaneous injection
  * Ribavirin in a dose of 13 mg/kg/day orally
  * Xerovirinc® 500mg twice daily orally.
  Interventions: Biological: Reiferon Retard in Arm 1; Drug: Bon one in Arm 3; Drug: Xerovirinc in Arm 2; Drug: Ribavirin in Arm 1

INTERVENTIONS:
Biological: Reiferon Retard in Arm 1 — Arm 1,2,3 Reiferon Retard® 160 µg /week subcutaneous injection for 48 weeks
  Other Names: Pegylated interferon alfa-2a (Reiferon Retard 160 µg ®)
Drug: Bon one in Arm 3 — Arm 3 , Bon One ® 0.5 µg daily orally for 48 weeks
  Arms: Arm 3 ( Bon one )
Drug: Xerovirinc in Arm 2 — Arm 2,3 Xerovirinc® 500mg twice daily orally for 48 weeks
  Other Names: Nitazoxanide
  Arms: Arm 2 ( Xerovirinc); Arm 3 ( Bon one )
Drug: Ribavirin in Arm 1 — Arm 1,2,3 Ribavirin in a dose of 13 mg/kg/day orally for 48 weeks

SUMMARY:
A single Center, Prospective Phase IV, Open-Label, Controlled, Randomized Trial comparing the efficacy, safety, and tolerability of Quadritherapy regimen (Reiferon Retard® , Ribavirin , Nitazoxanide and Alfacalcidol (Bon-One ® ) versus Triple therapy regimen (Reiferon Retard® , Ribavirin and Nitazoxanide) versus the standard of care regimen(Reiferon Retard® and Ribavirin) in the treatment of Naïve chronic hepatitis C among the Egyptian population. Effectiveness will be evaluated based on Sustained Virological Response (SVR) .

PRIMARY OBJECTIVE(S): The primary objectives of this trial are as follows:

* To compare the efficacy of the three treatment arms in naïve Chronic Hepatitis C Virus (HCV) genotype 4 patients by evaluating the sustained virological response ( SVR) at week 60 ( 3 months after end of treatment period)
* Identify optimum treatment protocol for HCV genotype 4 in respect to used combination of medications
* Whether adding vitamin D, a potent immunomodulator, could improve viral response.

STUDY DESIGN: This is a phase IV, single center, open labeled, randomized (1:1:1) controlled study.

NUMBER OF EVALUABLE SUBJECTS: 300 NUMBER OF CENTER/S: 1 Country:Egypt DURATION OF THE STUDY: 94 weeks TREATMENT: randomized 1:1:1 ratio into 3 Arms SUBJECT POPULATION: male or female subjects assessed by BMI less than 35, between the ages of 20 and 50 years. Subjects have to be diagnosed as Naïve Chronic Hepatitis C genotype 4 patients with compensated liver disease assessed by hematological and biochemical tests.

- DURATION OF THE STUDY: 94 weeks as follows:

Estimated Enrollment Duration: 16 weeks Collection of last Case Report Form (CRF) : 2 weeks from Last patient out. Queries Resolution: 4 weeks from Collection of last CRF. Database lock planned date: 2 weeks from Quires resolution. Final Study Report: 8 weeks from Database lock. Estimated duration of subject participation: 62 weeks as follows;

* Screening period per subject = 2 weeks
* Treatment phase per subject = 48 weeks
* Follow-up phase per subject = 12 weeks

N.B : Each patient will receive medications for Maximum 48 weeks if his/her Polymerase Chain Reaction (PCR) -ve at weeks 12 and 24 , and if his/her PCR +ve at week 12 or week 24 the treatment will be stopped .

ELIGIBILITY:
Inclusion Criteria:

1. The subject signs and dates a written informed consent form (ICF) prior to any study-related activities, including discontinuation of any prohibited medications.
2. If the subject is male and sexually active, he is eligible to enter and participate in this study if his partner(s) meet the criteria outlined in 2a or if he or his partner(s) are using one of the methods of birth control outlined in 2b. If the subject is female, she is eligible to enter and participate in this study if she meets the following criteria:

   1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is postmenopausal; for purposes of this study, postmenopausal is defined as 1 year without menses); or
   2. Childbearing potential, has a negative serum pregnancy test at screening.
3. The subject is between the ages of 20 and 50, inclusive at the time of the screening visit.
4. The subject is an ambulatory outpatient. Ambulatory is defined as not depending exclusively on a wheelchair for mobility. Nursing home subjects may be enrolled provided they are ambulatory. Subjects with spinal cord injuries resulting in paraplegia may not be enrolled.
5. The subject is or has been diagnosed with Hepatitis C genotype 4.
6. Subjects are treatment Naive
7. Male or female subjects with BMI ≤ 35 .
8. Compensated liver disease with all the following minimum hematological and biochemical criteria:

   1. Hemoglobin > 12 g/dl for males, >11 g/dl for females.
   2. White blood cell count (WBC) > 3,000 /mm3 - Absolute Neutrophilic count (ANC above 1000)
   3. Platelets > 80,000/mm3
   4. Prothrombin time less than 4 seconds above the upper limit of normal (ULN).
   5. Serum albumin > 3.5mg/dl
   6. Normal Bilirubin level (except for Gilbert's syndrome where indirect Bilirubin should be < 3mg/dl)
   7. Histological diagnosis of chronic hepatitis with Fibroscan( fibrosis assessment).
   8. Normal fasting blood glucose level or within 20% of ULN for non-diabetic patients. If there is a history of diabetes, hemoglobin A1C <8.5% (as evidence of good glucose control in recent months).
9. Serum Creatinine within normal limits.
10. Thyroid Stimulating Hormone (TSH) within normal limits of testing lab. Patients requiring medications to maintain TSH are eligible if they have fulfilled all other inclusion and exclusion criteria.
11. Alpha Fetoprotein within normal range obtained during one year prior to entry in the study. Results above the upper limit of normal but less than 100 units require both of the following:

    1. Alpha Fetoprotein obtained within 3 months of entry.
    2. Abdominal Ultrasound within 3 months of entry that is negative for evidence of hepatocellular carcinoma.
    3. If Alpha Fetoprotein is above 100 units CT scan of the abdomen that is negative for evidence of hepatocellular carcinoma is required.
12. Patients must be serum hepatitis B surface antigen (HBsAg) negative.
13. Negative Antinuclear Antibodies (ANA) or titer of < 1:160
14. Serum positive for anti-HCV antibodies and HCV-RNA.
15. Abdominal Ultrasound obtained within one year prior to entry in the study
16. Electrocardiogram for men aged > 40 years.
17. Normal urine analysis.
18. Normal fundus exam.
19. Serum Schistosoma antibody test, if positive > 1/80, a rectal biopsy is required. If rectal biopsy is positive to living Schistosomal eggs, treatment of Active Schistosomal disease is required one month prior to enrollment.

Exclusion Criteria:

1. The subject has been diagnosed with HBV or HCV of any genotype other than genotype 4 and /or HIV.
2. Subjects are older than 50 years or younger than 20 years of age.
3. Women who are pregnant or breast-feeding.
4. Suspected hypersensitivity to Interferon or Ribavirin.
5. Subjects with organ transplant other than corneal or hair transplant.
6. Any cause of the liver disease based on the patient's history and biopsy other than chronic hepatitis C genotype 4, including but not limited to:

   1. Alpha 1-antitrypsin deficiency.
   2. Wilson's disease.
   3. Liver transplant patients.
   4. Autoimmune hepatitis.
   5. Alcoholic liver disease.
   6. Obesity induced disease.
   7. Drug related liver disease.
   8. Co-infection with Hepatitis B Virus (HBV) or HIV (HBsAg or HIV antibodies positivity).
   9. Hemochromatosis (iron deposition more than 2+ in liver parenchyma)
   10. Evidence of advanced liver disease such as history or presence of ascitis, bleeding varices, spontaneous encephalopathy.
7. In the opinion of the investigator, the subject has a concurrent illness or disability (excluding HCV genotype 4) that may affect the interpretation of clinical efficacy and/or safety data or otherwise contraindicates participation in this clinical study ;

   1. Unstable pulmonary, endocrine & metabolic disorders e.g. poorly controlled diabetes.
   2. Subjects with hemophilia or any hemoglobinopathy including but not limited to thalassemia major or minor.
   3. Bone marrow compromise contraindicated for interferon treatment
   4. Central Nervous System (CNS) trauma or active seizures that require medications.
   5. The subject exhibits renal impairment as evidenced by a serum Creatinine higher than 2.0 mg/dL. Or history of Chronic renal failure
   6. Immunologically mediated diseases (e.g. inflammatory bowel disease, idiopathic thrombocytopenic purpura, systemic lupus erythromatosis, autoimmune hemolytic anemia, scleroderma, severe psoriasis, clinical cryoglobulinemia)
   7. Any medical condition requiring or likely to require during course of the study, chronic systemic administration of steroids.
   8. Patients with clinically significant retinal abnormalities.
   9. The subject has a history of unstable or deteriorating cardiac disease within the previous 6 months, including, but not limited to, the following:

   i. Myocardial infarction, unstable angina pectoris, coronary artery bypass surgery, or coronary angioplasty ii. Congestive heart failure requiring hospitalization iii. Uncontrolled arrhythmias
8. The subject has been diagnosed with a major psychiatric disorder (e.g., major depression or psychoses) within the past 2 years that required hospitalization and/or involved an attempted suicide. Subjects diagnosed with a major psychiatric disorder that did not require hospitalization or involve an attempted suicide must have remained on a stable dose of medication for at least 6 months prior to the screening visit.
9. The subject has a history of alcohol or substance abuse within the past 2 years.
10. The subject has a positive stool sample for ova or parasite (exception: the finding of Entamoeba coli is not exclusionary).
11. The subject has any evidence or treatment of malignancy (other than localized basal cell cancer, squamous cell skin cancer, or cancer in situ that has been resected) within the previous 5 years.
12. The subject used an investigational drug or participated in an investigational study within 30 days of screening.
13. The subject refuses to discontinue one (or more) prohibited medications at least 7 days prior to the screening visit.
14. The subject refuses to maintain a stable dose of one (or more) allowable concurrent medications for at least 30 days prior to the screening visit.
15. The subject is unable or unwilling to follow directions.
16. Contraindications to ribavirin and thus combination therapy include marked anemia, renal dysfunction, and coronary artery or cerebrovascular disease, and inability to practice birth control.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-01 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Early virological response | 3 months after start of treatment
  Early Virological Response (EVR) achieved by undetected Hepatitis C Virus (HCV) RNA after 12 weeks ( 3 months after start of treatment)

SECONDARY OUTCOMES:
Sustained Virological Response ( SVR ) | 3 months after end of treatmet ( Week 60)
  Sustained Virological Response ( SVR ) achieved by undetected HCV RNA after 1 year and 12 weeks (3 months after end of treatment) .

OTHER OUTCOMES:
Safety outcome | During the period of study medications taking (up to 48 weeks)
  Any adverse event will be found during the period of study medications taking will be recorded .

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Esmat, MD, Principal Investigator — Cairo University; Rasha Ahmed, MD, Study Director — Cairo University
Locations (1):
- Faculty of Medicine , Cairo University, Cairo, Cairo Governorate, Egypt